CLINICAL TRIAL: NCT01619644
Title: Rubinstein-Taybi Syndrome: Functional Imaging and Therapeutic Trial
Acronym: RUBIVAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Fondation Syndrome de Rubinstein-Taybi (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHUBX 2011/20
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Rubinstein-Taybi Syndrome
Keywords: RTS; Rubinstein Taybi; explorative phase 2; clinical approach; biological approach; motor skills
MeSH Terms: conditions — Rubinstein-Taybi Syndrome | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Valproate (Experimental): Group of 40 patients receiving one year of sodium valproate
  Interventions: Drug: sodium valproate
- Placebo (Placebo Comparator): Group of 20 patients receiving one year of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sodium valproate — sodium valproate (HDAC inhibitor) with an oral dosage of 30 mg/kg/jour
  Arms: Sodium Valproate
Drug: Placebo — Placebo with an oral dosage of 30 mg/kg/jour
  Arms: Placebo

SUMMARY:
An exploratory phase 2 therapeutic trial in children from 6 to 21, RTS carriers, randomized to be treated either with sodium valproate with the usual pediatric dosage (30 mg/kg/j), or by placebo for one year.

The investigator would like to include children because they could best profit from it due to their neuronal plasticity as CBP and EP300 take effect through neuronal and synaptic plasticity.

The therapeutic effect of sodium valproate in RTS patients will be assessed thanks to a clinical approach (learning and memory neuropsychological evaluation, fine motor skills assessment by pointing), to a biological approach (histone acetylation functional tests), and to imaging (morphological and functional MRI).

DETAILED DESCRIPTION:
Such a multidisciplinary approach has never been presented for this syndrome; it should enable us identifying specific cognitive and motor deficits and their association thanks to imaging markers. Assessing the various aspects of motor skills, i.e. primary (movements, standing at ease position, immobility) and complex motor skills (actions and behaviours, motor aspects of feelings and language expressions) is an integral part of the clinical examination in psychiatrics.

The main interest of a functional capacity analysis is to be used as an index allowing the assessment of the nervous system's global capacities and the study of the connections between cognitive functions and motor skills Main objective: Evaluate long term memory with subtest "point location" - CMS and "image recognition" RBMT A patient is said to be responder if after one year his or her test result increase for one point at least one of the two tests : a increase of one point to "point location" or "image recognition".

Double-blind phase 2 clinical trial, designed as a one-step Fleming design but with a control group. Rubival is a two-parallel group randomized trial:

* a placebo group of 20 patients
* a group of 40 patients taking sodium valproate (HDAC inhibitor) with an oral dosage of 30 mg/kg/jour

ELIGIBILITY:
Inclusion Criteria:

* Children over 6 and under 21
* RTS confirmed by a genetic study with a CBP gene or EP300 gene mutation
* Sufficient cognitive capacities for neuropsychological evaluation
* Free and informed consent of the parents or guardians
* Children affiliated to or benefiting of the French social welfare system

Exclusion Criteria:

* Contraindication to sodium valproate
* Women of reproductive age without effective contraception means
* Case history of sodium valproate treatment
* Monotherapy treatment for epilepsy with Lamictal with a dosage superior to 5 mg/kg/j
* Family history of severe hepatitis including drug
* Acute or chronic hepatitis
* Pregnancy

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2012-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Memory tests (assessing memory learning) | 1 year
  The main outcome measure was to evaluate long term memory with two subtests :
  * point location, subtest of CMS (children memory scale). The score ranges from 0 to 6
  * image recognition, subtest of RBMT (Rivermead Behavioural Memory Test). The score range from 0 to 10. One point for each image recognized A patient is said to be responder if after one year of treatment , his or her test result increase for one point at least one of the two tests

SECONDARY OUTCOMES:
Special brain imaging profile and motor skills (posturology and motor coordination in a visio-manual pointing task) | 1 year
  For motor skills, the profile was based on 3 tasks : posturology, motor coordination in a visuo-manual pointing task and in mobile interception task..
  For brain imaging, a variety of outcome measures will be used for example, brain volume, anisotropy fraction, diffusion coefficient for structural magnetic imaging and the signal intensity for functional Magnetic Resonance Imaging
Cognitive and developmental profile | 1 year
  Based on the results of several battery test and evaluation scale, VABS II (Vineland Adaptative Behaviour Scale II), Leiter R, EVIP, ECOSSE, NEPSY : fluency verbal sutest, CMS : 2 subtests, RBMT : 1 subtest
Histone acetylation profile | 1 year
Global acetylation level | 1 year
Acetylation level of selected gene | 1 year
Measurement of selected gene expression | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Didier LACOMBE, PU-PH, Principal Investigator — University Hospital Bordeaux, France; Paul PEREZ, PH, Study Chair — University Hospital Bordeaux, France
Locations (1):
- University Hospital Bordeaux, France, Bordeaux, France